CLINICAL TRIAL: NCT00906321
Title: Facilitating Web-Based Patient Decision Support: Decision About Medication to Lower Breast Cancer Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 999909150; 09-C-N150; NCT00953238 (obsolete NCT alias)
Record Dates: First submitted 2009-05-20; First posted 2009-05-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-05-26

CONDITIONS: High Risk for Breast Cancer; Risk Reduction Behavior
Keywords: Web-Based Decision Support; Breast Cancer Risk
MeSH Terms: conditions — Risk Reduction Behavior

INTERVENTIONS:
Behavioral: Web-Based Decision Support

SUMMARY:
Background:

* Chemoprevention is the use of preventive medications to reduce the risk of breast cancer for women who are at a high risk of developing the disease. Although the treatment has shown effectiveness in preventing cancer development, chemoprevention is notably underutilized even by women who are at a high risk of developing breast cancer.
* Researchers are interested in determining if better decision support mechanisms, such as interactive Web sites, can help to overcome some of the barriers to chemoprevention.

Objectives:

- To develop and test a prototype Web-based module that will provide decision support to women who are considering chemoprevention for breast cancer.

Eligibility:

* Women 35 years of age and older who are at high risk for breast cancer and whose doctor has recommended chemoprevention (either Tamoxifen or Raloxifene), and who have no other history of cancer (apart from non-melanoma skin cancer or precancerous cervical lesions).
* Participants must have a working e-mail address and access to a computer with internet access and a telephone.

Design:

* Participants who are considering chemoprevention will be randomized to a Web-based decision support module or standard care online information resources.
* Participation lasts two months and involves using the online resources provided and filling out questionnaires two times during the study (at the beginning and the end).

The first time will be at the begin of the study.

* No medical treatments are offered as a part of this study

DETAILED DESCRIPTION:
BACKGROUND:

* Breast cancer chemoprevention has been notably underutilized.
* Barriers to integrating breast cancer risk reducing measures include: lack of time, low priority of risk reduction in comparison to treatment, the need to personalize risks and benefits of chemoprevention, and the need for resources/information necessary for women to make informed decisions.
* Access to quality decision support resources to facilitate making informed, preference-sensitive decisions about chemoprevention may provide a mechanism to overcome some of the current barriers to chemoprevention utilization.

OBJECTIVES:

* Develop and refine a web-based patient decision support module for high-risk women making a decision about breast cancer chemoprevention.
* Conduct a randomized study of TACHD decision support versus standard care online information support to evaluate the impact of the chemoprevention module of the TACHD decision support intervention.

ELIGIBILITY:

* Women with no history of cancer other than cervical carcinoma in situ or non-melanoma skin cancer
* High risk for breast cancer based on at least one of the following:

  * Gail score > 1.67
  * History of atypical hyperplasia (either ductal or lobular)
  * History of lobular carcinoma in situ
  * Documentation of a deleterious BRCA1 or BRCA2 mutation
* Considering a decision about chemoprevention with tamoxifen or raloxifene
* Access to an IBM-compatible or MacIntosh personal computer with broadband Internet access
* Access to an email account
* Access to a telephone
* Aged 35 or older
* Able to communicate in English verbally and in writing

DESIGN:

* The project will be guided by the Cognitive-Social Health Information Processing (CSHIP) model overall, and incorporate the Ottawa Decision Support. Framework (ODSF) in one consistent decision support process.
* Testing of the chemoprevention decision support module will be conducted in a two-group pre- post-test experimental design with 64 at-risk women identified through Fox Chase Risk Assessment Programs and the NCI Clinical Cancer Genetics Program (CCGP) at the National Naval Medical Center (NNMC).
* A process evaluation analysis will assess participants' experiences using TACHD.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Women with no history of cancer other than cervical carcinoma in situ or non-melanoma skin cancer
2. High risk for breast cancer based on at least one of the following:

   * Gail score > 1.67
   * History of atypical hyperplasia (either ductal or lobular)
   * History of lobular carcinoma in situ
   * Documentation of a deleterious BRCA1 or BRCA2 mutation
3. Considering a decision about chemoprevention with tamoxifen or raloxifene
4. Access to an IBM-compatible or MacIntosh personal computer with broadband Internet access
5. Access to an email account
6. Access to a telephone
7. Aged 35 or older
8. Able to communicate in English verbally and in writing
9. Women of all races and ethnic groups are eligible for this study.

EXCLUSION CRITERIA:

1. Concurrent participation in another cancer chemoprevention study
2. Prior history of cancer, other than cervical carcinoma in situ or non-melanoma skin cancer
3. Ever taken tamoxifen or raloxifene
4. Age less than 35
5. Unable to communicate in English verbally and in writing
6. No computer with internet access
7. No email account
8. No telephone

Ages: 35 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2009-05-18; Primary Completion 2010-05-26 (Actual); Study Completion 2010-05-26 (Actual)

PRIMARY OUTCOMES:
Conduct a formative evaluation of the impact of the chemoprevention module of the Trusted Advisor for Cancer Health Decisions (TACHD) decision support intervention

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Guttmacher AE, Collins FS. Genomic medicine--a primer. N Engl J Med. 2002 Nov 7;347(19):1512-20. doi: 10.1056/NEJMra012240. No abstract available. PMID 12421895
- [Background] Collins FS. Shattuck lecture--medical and societal consequences of the Human Genome Project. N Engl J Med. 1999 Jul 1;341(1):28-37. doi: 10.1056/NEJM199907013410106. No abstract available. PMID 10387940
- [Background] Rose AL, Peters N, Shea JA, Armstrong K. Attitudes and misconceptions about predictive genetic testing for cancer risk. Community Genet. 2005;8(3):145-51. doi: 10.1159/000086757. PMID 16113531